CLINICAL TRIAL: NCT04480580
Title: Seroprevalence of SARS-Cov-2 in the Setting of a Non-dedicated COVID-19 Hospital in a Low CoV-2 Incidence Area: Implications for Surgery
Status: Completed | Type: Observational
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Fabio Medas, Assistant Professor, University of Cagliari
Other Study IDs: COVID-SURG
Record Dates: First submitted 2020-07-20; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Covid19; Surgery; SARS (Severe Acute Respiratory Syndrome)
Keywords: SARS-CoV-2, surgery
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized patients
  Interventions: Diagnostic Test: SARS-CoV-2 Ab

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 Ab — Patient test for specific antibodies for SARS-CoV-2

SUMMARY:
We have herein analysed the patients admitted to our Department that underwent serologic tests for SARS-CoV-2 either by Ab or RT PCR, to estimate the prevalence of COVID-19 in the setting of a non-dedicated COVID-19 hospital and in a low CoV-2 incidence area, and to evaluate if security measures are necessary for this context.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized during pandemic spread

Exclusion Criteria:

* Incomplete data

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in surgical department
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Seroprevalence of SARS-CoV-2 | 3 months
  Positivity of specific IgM or IgG

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Cagliari, Cagliari, CA, Italy

IPD SHARING:
Plan to Share IPD: No